CLINICAL TRIAL: NCT06345365
Title: A Prospective, Multicenter, Randomized Controlled Study on the MA+AZA Regimen for the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: MA+AZA Regimen for the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanxi Province Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Jingzhou Central Hospital (Other); Yichang Central People's Hospital (Other); Taihe Hospital (Other); Central Hospital of Xiaogan (Other); Xianning Central Hospital (Other); The First People's Hospital of Jingzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09
Record Dates: First submitted 2024-02-01; First posted 2024-04-03 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Mitoxantrone liposome; Newly diagnosed AML patients; Ara-Cytarabine; Azacytidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mitoxantrone liposome, Ara-Cytarabine and azacitidine (Experimental): Mitoxantrone hydrochloride liposome 24 mg/m2, IV every 4 weeks, day 1; Ara-Cytarabine 100 mg/m2, IV every 12 h, days 1-7; Azacitidine 100 mg, subcutaneous, once daily, days 1 to 7;
  Interventions: Drug: mitoxantrone liposome, Ara-Cytarabine and azacitidine
- Daunorubicin, Ara-Cytarabine and azacitidine (Active Comparator): Daunorubicin 60 mg/m2, intravenously, once daily, days 1 to 3 Ara-Cytarabine 100 mg/m2, IV drip, every 12h, days 1 to 7; Azacitidine 100 mg, subcutaneous, once daily, days 1 to 7;
  Interventions: Drug: Daunorubicin,Ara-Cytarabine, azacitidine

INTERVENTIONS:
Drug: mitoxantrone liposome, Ara-Cytarabine and azacitidine — Mitoxantrone hydrochloride liposome 24 mg/m2, IV every 4 weeks, day 1; Ara-Cytarabine 100 mg/m2, IV every 12 h, days 1-7; Azacitidine 100 mg, subcutaneous, once daily, days 1 to 7
  Arms: mitoxantrone liposome, Ara-Cytarabine and azacitidine
Drug: Daunorubicin,Ara-Cytarabine, azacitidine — Daunorubicin 60 mg/m2, intravenously, once daily, days 1 to 3; Ara-Cytarabine 100 mg/m2, IV drip, every 12h, days 1 to 7; Azacitidine 100 mg, subcutaneous, once daily, days 1 to 7;
  Arms: Daunorubicin, Ara-Cytarabine and azacitidine

SUMMARY:
Investigator proposed to apply the new dosage form of mitoxantrone hydrochloride liposomes to the clinical treatment of AML, while combining with cytarabine and azacitidine to form the MA+AZA treatment regimen(Mitoxantrone liposome +Ara-Cytarabine+Azacitidine), which would provide an optimal induction treatment regimen for patients with primary AML by comparing with the traditional chemotherapy regimen, DA+AZA (Daunorubicin+Ara-Cytarabine+Azacitidine).

DETAILED DESCRIPTION:
In this study, AML patients were randomly divided into MA+AZA treatment group and DA+AZA treatment group by conducting a prospective, multicentre, exploratory, randomised controlled study. By observing the efficacy and safety of the MA+AZA combination regimen in the treatment of primary AML, and comparing the superiority of the traditional regimen, high-quality clinical evidence was obtained, providing practical evidence to support the improvement of the intervention effect and clinical prognosis of primary AML.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary AML with morphologically and immunologically confirmed diagnosis of bone marrow;
2. Age 18-75 years old;
3. Liver and renal function: serum total bilirubin ≤1.5 × upper limit of normal (ULN), AST/ALT <2 × ULN, serum creatinine <1.5 × ULN, 80 ml/min ≤ creatinine clearance ≤120 ml/min;
4. Cardiac function: ejection fraction EF ≥50%, ultrasensitive troponin and natriuretic peptide <1.5 × ULN;
5. Physical condition: ECOG score 0-2;
6. Obtained informed consent signed by the patient or family.

Exclusion Criteria:

1. Allergy or significant contraindication to any of the drugs involved in the protocol;
2. Patients with concomitant myelofibrosis;
3. Severe cardiac disease, including myocardial infarction and cardiac insufficiency;
4. Concomitant malignant tumours of other organs;
5. Patients with active tuberculosis and HIV-positive patients;
6. Other blood system diseases at the same time;
7. Pregnant or breastfeeding women;
8. Inability to understand or comply with the study protocol;
9. Previous intolerance or allergy to similar drugs;
10. Concurrent participation in other clinical studies;
11. Any other condition that prevents the study from proceeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | Efficacy evaluation at 2-3 weeks after the first cycle (each cycle is 28 days)
  Bone marrow primitive cells <5%, no primitive cells with Auer vesicles, no primitive cells in the peripheral blood, no extramedullary leukaemia, neutrophil count ≥1.0×109/L, platelet count ≥100×109/L.

SECONDARY OUTCOMES:
Incidence of adverse events | Efficacy evaluation at 2-3 weeks after the first cycle (each cycle is 28 days)
  Incidence of adverse events, e.g., GI adverse reactions, cardiotoxicity, etc.
Compound CR rate | Efficacy evaluation at 2-3 weeks after the first cycle (each cycle is 28 days)
  CR+ CRi
Objective remission rate | Efficacy evaluation at 2-3 weeks after the first cycle (each cycle is 28 days)
  CR+CRi+MLFS+PR
No remission rate | Efficacy evaluation at 2-3 weeks after the first cycle (each cycle is 28 days)
  Patients not meeting criteria for CR, CRi, MLFS or PR
Event-free survival | Assessment of up to 100 months from the date of randomisation to the date of first recorded progress or the date of death from any caus)
  From the date of the patient's first dose to the date of treatment failure,haematological relapse after CR/CRi or all-cause mortality, whichever occurs first
Disease-free survival | From date of achieving remission to date of relapse or death from any cause (Assessment of up to 100 months from the date of randomisation to the date of first recorded progress or the date of death from any cause, whichever comes first)
  For patients achieving CR or CRi only, from the date of achieving remission to the date of relapse or death from any cause
Overall survival | Time from the patient's first dose of medication to death from any cause (Assessment of up to 100 months from the date of randomisation to the date of first recorded progress or the date of death from any cause, whichever comes first)
  The time from the patient's first dose of medication to the time of death from any cause.
Mortality rate | 30 days, 60 days after starting treatment; Assessment of up to 100 months from the date of randomisation to the date of first recorded progress or the date of death from any cause, whichever comes first
  Early deaths: all-cause deaths within the timeframe associated with study treatment (e.g., 30 days, 60 days after starting treatment); Cumulative deaths: deaths within the period from the date of achieving remission to the date of no prior relapse for patients achieving CR or CRi only.

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Zhou, Study Director — Wuhan University
Locations (11):
- China (11):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Central Hospital of Huanggang, Huanggang, Hubei
  - The First People's Hospital of Jingzhou, Jingzhou, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Shiyan Taihe Hospital, Shiyan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - The Central Hospital of Xiaogan, Xiaogan, Hubei
  - Yichang Central Hospital, Yichang, Hubei
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Wuxi, Jiangsu
  - Shanxi Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No